CLINICAL TRIAL: NCT02187718
Title: A Prospective Single-centre Randomised Controlled Clinical Trial Comparing Sentinel Node Procedure Under Local Anaesthesia to Traditional Sentinel Node Procedure Under General Anaesthesia in Patients <60 Years With a Breast Carcinoma >20 mm.
Brief Title: Ambulatory SNP Under Local Anaesthesia in a Subgroup of Breast Cancer Patients - Trial
Acronym: AMBULANT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Medical Center Alkmaar (Other)
Responsible Party: Principal Investigator, M.W.H. Leenders, M.W.H. Leenders, M.D., Medical Center Alkmaar
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: NL49489.094.14
Record Dates: First submitted 2014-07-09; First posted 2014-07-11 (Estimated); Last update posted 2014-07-11 (Estimated); Status verified 2014-07

CONDITIONS: Breast Neoplasms
Keywords: Sentinel Lymph Node Biopsy; Local Anaesthesia
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- SNPGA (Other): Sentinel Node Procedure under General Anaesthesia
  Interventions: Procedure: Sentinel Node Procedure under General Anaesthesia
- SNPLA (Other): Sentinel Node Procedure under Local Anaesthesia
  Interventions: Procedure: Sentinel Node Procedure under Local Anaesthesia

INTERVENTIONS:
Procedure: Sentinel Node Procedure under Local Anaesthesia
  Arms: SNPLA
Procedure: Sentinel Node Procedure under General Anaesthesia
  Arms: SNPGA

SUMMARY:
Rationale: In breast cancer (BC) patients, lymph node status is a key prognostic indicator. At present, axillary ultrasound (US) with subsequent fine needle aspiration cytology (FNAC) of suspicious lymph nodes (US+FNAC) is widely used as a pre-operative staging method. When US+FNAC is negative, a sentinel node procedure (SNP) is performed during breast surgery. Nowadays, an axillary lymph node dissection (ALND) is generally performed if one of the abovementioned diagnostic entities reveals lymph node metastases. However, the extensive role of ALND in BC patients with lymph node metastases may change or diminish in upcoming years due to emerging evidence that completion ALND (cALND) does not affect disease-free survival and overall survival in early BC patients with (sentinel) node-positive disease. Whether ALND is needed in these patients, should be based on (axillary) tumour load. Because of the fact that tumour load can only be reliably evaluated by SNP and not by US+FNAC, the role of SNP might become even more important in upcoming years.

Ideally, the status of this sentinel lymph node is known prior to breast surgery, so a patient tailored treatment plan can be made and discussed with the patient before breast surgery. In this context, it would be very logical to perform a SNP under local anaesthesia (LA), prior to breast surgery. This might not only lead to significantly less two-step surgical procedures under general anaesthesia (GA), but might also lead to a reduction of depressive symptoms and anxiety and improved quality of life (QoL) of BC patients, because BC patients are in particular risk for psychological distress in the first three months after diagnosis of BC. Knowing lymph node status and the complete treatment plan as soon as possible (by performing a SNP under LA), might reduce this psychological distress. To investigate which BC patients would benefit most from SNP under LA, the investigators recently analysed 1132 BC patients retrospectively. Both prevalence of axillary lymph node metastases and prevalence of false negative results of US+FNAC were directly associated with age <60 years and with primary breast tumour size >20 mm. Hence, these BC patients might benefit most from SNP under LA. In the present study, the value of SNP under LA in these BC patients (i.e. <60 years with a breast carcinoma >20 mm) will be analysed.

Objectives: Reduction of the mean number of operations under general anaesthesia per patient. Improvement of QoL. Reduction of depressive symptoms and experienced anxiety.

Study design: Prospective single centre randomised controlled clinical trial. Study population: Women aged 18 to 60 years who are diagnosed with BC AND with a tumour size of >20 mm ultrasonographically AND with a negative or inconclusive pre-operative US+FNAC.

Intervention: Sentinel Node Procedure under Local Anaesthesia (SNP under LA) Control: Traditional Sentinel Node Procedure under General Anaesthesia (SNP under GA) Main study parameters: Primary outcome parameters are the number of operations under GA per patient and the number of operations under LA per patient. Secondary outcome parameters are QoL, experienced depressive symptoms and anxiety.

Timeline and statistics: The inclusion period will be conducted from the 1st of July 2014 to the 1st of August 2015, and 80 patients will be enrolled in this study (alpha 0.05; power 0.8). Inclusion of 80 patients will be sufficient to reduce the number of two-stage surgical procedures under general anaesthesia with 30%. Data will be analysed using descriptive statistics, Chi-squared test, Fisher's exact test, Mann-Whitney U test, Kruskall-Wallis test, students t-test, ANOVA, paired t-test, Wilcoxon signed-rank test, Friedman test, Pearson's and Spearman's rank correlation coefficients and finally logistic and linear regression analysis.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age 18-60 years
* Diagnosis of invasive BC (established with core needle biopsy of the breast lesion)
* Breast carcinoma measures > 20 mm ultrasonographically
* Pre-operative US+FNAC is negative or inconclusive
* No evidence of distant metastases
* ASA Classification I-III
* Signed informed consent

Exclusion Criteria:

* History of previous breast surgery in the affected breast
* History of previous axillary surgery in the ipsilateral axilla
* History of radiation therapy (ipsilateral breast or axilla)
* History of neo-adjuvant therapy (for the BC)
* Known allergy to lidocain

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2015-01; Primary Completion 2016-12 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Number of operations under general anaesthesia | 6 months
Number of operations under local anaesthesia | 6 months
The number of patients in whom breast surgery is performed ≤21 days. | 6 months

SECONDARY OUTCOMES:
Quality of Life | 6 months
  Quality of Life is measured with the WHOQOL-bref questionnaire
Depressive symptoms | 6 months
  Depressive symptoms are measured with the Centre for Epidemiological Studies-Depression scale (CES-D)
Anxiety | 6 months
  Anxiety is measured with the State-and-Trait-Anxiety-Inventory (STAI)

OTHER OUTCOMES:
Pain during SNP under local anaesthesia | 6 months
  Pain during SNP under local anaesthesia is measured with a Numeric Pain Rating Scale
Duration of SNP under local anaesthesia | 6 months
Duration of SNP under general anaesthesia | 6 months
Number of lymph nodes excised by SNP under local anaesthesia | 6 months
Number of lymph nodes excised by SNP under general anaesthesia | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Hermien Schreurs, MD, PhD, Principal Investigator — Medical Center Alkmaar
Locations (1):
- Medical Center Alkmaar, Alkmaar, North Holland, Netherlands